CLINICAL TRIAL: NCT06302205
Title: A Home-based Exercise and Physical Activity Intervention After Liver Transplantation: Impact of Exercise Intensity - a Monocenter Randomized Controlled Trial [PHOENIX-Liver]
Brief Title: A Home-based Exercise and Physical Activity Intervention After Liver Transplantation: Impact of Exercise Intensity
Acronym: PHOENIX-L
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S66232
Record Dates: First submitted 2023-12-06; First posted 2024-03-08 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-11

CONDITIONS: Liver Transplantation; Physical Fitness
Keywords: Exercise Intensity
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two interventional groups and one control group
Who Masked: Outcomes Assessor
Masking Description: The nature of the intervention does not allow blinding of study participants. However, outcome assessors and data investigators will be blinded to the participants' group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham Group (Sham Comparator): Home-based low-intensity exercise training without subsequent physical activity intervention.
  Interventions: Other: Sham intervention
- Moderate-intensity (MIT) (Experimental): Home-based moderate-intensity exercise training with subsequent physical activity intervention.
  Interventions: Other: Physical activity
- Combined moderate and high-intensity (MHIT) (Experimental): Home-based moderate- and high-intensity exercise training with subsequent physical activity intervention.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — The home-based training intervention consists of two phases of each three months in duration. It consists of three weekly aerobic training sessions on the one hand, and two weekly training sessions focused on strength, balance, and flexibility on the other hand.
  Arms: Combined moderate and high-intensity (MHIT); Moderate-intensity (MIT)
Other: Sham intervention — 2 times a week, flexibility and balance training
  Arms: Sham Group

SUMMARY:
Research demonstrated that transplant recipients benefit from physical activity, but there is a gap in knowledge regarding the required intensity. In the PHOENIX-Liver study, researchers aim to investigate the adequate intensity of rehabilitation programs after liver transplantation. Patients will be randomized into one of the three PHOENIX-Liver training groups (low, moderate, moderate to high). The six months rehabilitation program is conducted from the patient's home but supervised by a PHOENIX-investigator.

At baseline, after three months of rehabilitation and after six months of rehabilitation, a test moment takes place at which physical fitness, cardiovascular health, liver function, and body composition will be assessed. Questionnaires are taken monthly to survey well-being, safety, quality of life, physical activity, and cost-effectiveness.

To gather information on the potential for implementation in a real-world setting, a 15-month-long physical activity phase will start after the intervention phase. This entails a maintenance physical activity program tailored to the patients' preferences. A follow-up at UZ Leuven is planned at three and at 15 months where the same clinical evaluations will be conducted as during the test moments of the intervention phase.

DETAILED DESCRIPTION:
Liver transplantation constitutes the only curative treatment for patients with end-stage liver disease. Advances in the field have led to favourable short- and medium term (1-3 year) post-transplant survival rates, but improvement in long-term survival rates remains disappointing. Due to the immunosuppressive therapy, a sedentary lifestyle and a poor recovery of post-transplant physical fitness, the proportion of liver transplant recipients that develop a new-onset or a deteriorating unfavourable cardiovascular risk profile is alarmingly high, and cardiovascular disease is the leading cause of death in this population. By consequence, in order to improve long-term outcome after liver transplantation, prevention of cardiovascular disease should be prioritized. The investigators are convinced that the challenge of cardiovascular disease and lack of physical fitness in liver transplant recipients should and can be addressed by subjecting these patients to a structured physical rehabilitation program. The aim of this project is implement a structured, individually-tailored, home-based but supervised physical rehabilitation and maintenance program for de novo liver transplantation recipients, and to demonstrate the feasibility and safety of such approach as well as its efficacy to improve physical fitness. The program will consist of a 2-phase intervention of i) home-based exercise training (aerobic exercise training as well as strength, flexibility and stability exercises under in-person and subsequently remote guidance) and ii) an 15-month maintenance phase of physical activity. This program will be studied in an open-label randomized trial where the regimen will be compared with a regimen of standard of posttransplant care. In addition to the interventional arm, two different regimens of exercise training intensity will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* de novo adult liver transplant recipients with a transplant vintage of two to three months
* access to a home freezer (± -18°C)

Exclusion Criteria:

* Aberrant CPET (abnormal low cardiorespiratory fitness is not considered an exclusion criteria), unstable angina, life-threatening arrhythmias, uncontrolled hypertension/diabetes, HbA1c ≥ 9%, severe pulmonary disease (FEV1 < 50%), musculoskeletal disorders not allowing physical training on a cycle ergometer, or any other medical reasons by the physician considered to be a contraindication for moderate or high-intensity physical exercise
* multi-organ transplantation (exception: combined liver-kidney transplant is considered eligible for participation)
* ongoing treatment for malignancies
* unable to understand Dutch
* no access to smartphone and/or computer with internet access
* does not willing to except the general conditions of Coachbox. Preparticipation medical screening (cardiopulmonary exercise testing with 12-lead ECG + stratification of cardiovascular risk factors) will be performed by a cardiologist (Dr. Kaatje Goetschalckx at UZ Leuven).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | At 0, 3 and 6 months of the interventional rehabilitation programme and at 15 months after the end of the intervention
  Changes in peak oxygen uptake (mL O2·min-1·kg-1) assessed by cardiopulmonary exercise test

SECONDARY OUTCOMES:
Functional exercise capacitiy | At 0, 3 and 6 months of the interventional rehabilitation programme and 15 months after the end of the intervention
  six-minute walking test (m)
Hand grip strength | At 0, 3 and 6 months of the interventional rehabilitation programme and 15 months after the end of the intervention
  assessement by means of Jamar Hydraulic Hand Dynamometry (kg)
Knee-extensor strength | At 0, 3 and 6 months of the interventional rehabilitation programme and 15 months after the end of the intervention
  assessement by means of Biodex dynamometer (Nm)
Endothelial function | At 0, 3 and 6 months of the interventional rehabilitation programme and 15 months after the end of the intervention
  assessed via flow mediated dilation
Arterial stiffness | At 0, 3 and 6 months of the interventional rehabilitation programme and 15 months after the end of the intervention
  assessed via pulse wave velocity
Graft function | At 0 and after 21 months
  Transient elastography Fibroscan assessing liver stiffness
Occurence of adverse events | Monthly
  Safety is estimated by means of questionnaires
Motor fitness | At 0, 3 and 6 months of the interventional rehabilitation programme and 15 months after the end of the intervention
  Short Physical Performance Battery test
Blood pressure | At 0, 3 and 6 months of the interventional rehabilitation programme and 15 months after the end of the intervention
  Variation in blood pressure measured by means of automatic device (Omron M6) in fasted condition and without medication taken in
Blood profile | At 0, 3 and 6 months of the interventional rehabilitation programme, and at 3 and 15 months after the end of the intervention
  Blood is drawn when patient is in fasted condition and did not take their medication

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leunis S, Van Criekinge H, Vrancken L, Vandecruys M, Renier M, De Geest S, Bogaerts S, De Smet S, H Van Craenenbroeck A, Monbaliu D, Cornelissen V. Understanding participation of liver transplant recipients in an exercise intervention RCT: a cross-sectional study of barriers and motivators. BMC Sports Sci Med Rehabil. 2025 Nov 10;17(1):324. doi: 10.1186/s13102-025-01369-y. PMID 41214814
- [Derived] De Smet S, Leunis S, Van Criekinge H, Vandecruys M, Vrancken L, Renier M, Fieuws S, Goetschalckx K, Luyten J, Raes J, Bogaerts S, De Geest S, Van Craenenbroeck AH, Cornelissen V, Monbaliu D. Home-based exercise and PHysical activity maintenance interventiOn after livEr traNsplantation: Impact of eXercise intensity (PHOENIX-Liver). BMJ Open Sport Exerc Med. 2025 Mar 15;11(1):e002436. doi: 10.1136/bmjsem-2024-002436. eCollection 2025. PMID 40098918